CLINICAL TRIAL: NCT01435174
Title: Pharmacokinetics of Single-Dose Oral Ranolazine in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Bruce A. Mueller, Associate Dean of Academic Affairs, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-259-0123, HUM00051141
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: End-stage Renal Disease; Cardiovascular Disease
Keywords: ranolazine; end-stage renal disease; pharmacokinetics; cardiovascular disease
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranolazine (Experimental): End-stage renal disease patients receiving a single-dose of ranolazine and a concomitant hemodialysis session.
  Interventions: Drug: Ranolazine; Procedure: Pharmacokinetic Blood and Dialysate Sampling; Procedure: QT Interval

INTERVENTIONS:
Drug: Ranolazine — A single dose of two oral ranolazine extended release 500 mg tablets
  Other Names: Ranexa
Procedure: Pharmacokinetic Blood and Dialysate Sampling — Blood samples collected to assess ranolazine plasma and dialysate concentrations.
  Other Names: Ranexa; PK sampling
Procedure: QT Interval — Calculation of a QT interval will be performed throughout subject participation.
  Other Names: Ranexa; QT interval calculation

SUMMARY:
End-stage renal disease (ESRD) patients often develop cardiovascular complications, and cardiovascular disease is the leading cause of death in this population. Ranolazine's ability to treat angina without reducing heart rate or blood pressure makes it an important option for ESRD patients. The hemodialysis clearance of ranolazine is unknown. A single-dose pharmacokinetic study is needed to characterize ranolazine and its metabolites in ESRD patients on and off hemodialysis. Results of the proposed study will provide initial dosing estimates for a follow-up, multiple-dose pharmacokinetic study in this population.

ELIGIBILITY:
Inclusion Criteria:

* 18-74 years of age
* Within 50% of ideal body weight and greater than 40 kg
* Chronic kidney disease (CKD) stage 5 receiving maintenance hemodialysis for at least 3 months
* Native kidney estimated glomerular filtration rate(GFR) < 10 mL/min
* No concurrent illness or evidence of infection
* Able to give informed consent

Exclusion Criteria:

* QTc interval > 470 msec at echocardiogram (ECG) obtained within the last 6 months
* Concomitant QT-prolonging drugs, major P-gp inhibitors, and CYP3A4 inducers and inhibitors including: cyclosporine, rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, St. John's Wort, ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, saquinavir, quinidine, dofetilide, sotalol, amiodarone, erythromycin, thioridazine, ziprasidone, haloperidol, trimethoprim/sulfamethoxazole, ciprofloxacin, norfloxacin, levofloxacin, moxifloxacin
* Pre-study hemoglobin < 9.5 g/dL
* Plasma albumin < 2.5 g/dL
* Liver disease - exclude subjects with a Child Pugh score of C or higher
* Positive pregnancy test
* Breastfeeding
* Allergy to ranolazine
* Participating in another investigational study
* Hepatitis B infection due to dialysis isolation requirements
* Unstable blood pressure control
* Need for routine large fluid removal during dialysis (> 4L)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Mueller, PharmD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Scoville BA, Segal JH, Salama NN, Heung M, Bleske BE, Eyler RF, Mueller BA. Single dose oral ranolazine pharmacokinetics in patients receiving maintenance hemodialysis. Ren Fail. 2019 Nov;41(1):118-125. doi: 10.1080/0886022X.2019.1585371. PMID 30909832

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine
Started | 17
Completed | 8
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Patients 18 to 74 with chronic kidney disease stage 5 receiving 3 times weekly maintenance hemodialysis for at least 3 months were considered for study inclusion. Patients had to weigh >40 kilograms, be within 50-150% of their ideal body weight, have an eGFR of <10 mL/min, have no evidence of infection, and be able to give informed consent.
Arm/Group | Ranolazine
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 33 [20 to 63]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters of Ranolazine
Description: Peak Plasma Concentration (Cmax) with a 500 mg dose of ranolazine
Time Frame: At hours post-dose: 0, 2, 4, 8, 12, 15, 18, 20, 22, 23, 26, 30, 65
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Ranolazine
Number analyzed (Participants) | 8
mcg/mL | 0.65 (0.27)

ADVERSE EVENTS:
Arm/Group | Ranolazine
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=8)
Elevated Potassium with EKG Changes (Cardiac disorders) | 1 — High potassium was determined to be due to needing dialysis and unlikely related to the administration of ranolazine. The subject admitted to drinking more than usual (including fruit juice) and not following renal diet over the weekend.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No